CLINICAL TRIAL: NCT01466647
Title: A Phase I Pilot Study of the IGF-1R Inhibitor AXL1717 in Combination With Gemcitabine HCL and Carboplatin in Previously Untreated, Locally Advanced, or Metastatic Squamous Non-small-cell Lung Cancer
Brief Title: A Study of the IGF-1R Inhibitor AXL1717 in Combination With Gemcitabine HCL and Carboplatin to Treat Non-small-cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axelar AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXL004
Record Dates: First submitted 2011-10-21; First posted 2011-11-08 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — picropodophyllin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AXL1717 in combination with Gemcitabine HCL and Carboplatin (Other): AXL1717 in combination with Gemcitabine HCL and Carboplatin
  Interventions: Drug: AXL1717

INTERVENTIONS:
Drug: AXL1717 — A repeated BID treatment for 14 days, followed by a 7 day observation period for two treatment periods

SUMMARY:
This is a open single-center, explorative, Phase I pilot dose finding study including patients treated with AXL1717 in addition to standard chemotherapy of gemcitabine HCL and carboplatin.

DETAILED DESCRIPTION:
Open single-center, explorative, Phase I pilot study including patients treated with AXL1717 in addition to standard chemotherapy of gemcitabine HCL and carboplatin. Patients will be treated within the study for 2 treatment cycles of 3 weeks each. Survival data will be obtained. Tumor assessment will be conducted at baseline and then at the end of the study period. Concomitant supportive therapies will be allowed.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Histologically or cytologically confirmed diagnosis of locally advanced, or metastatic squamous non-small-cell lung cancer (stage IIIB or IV) and scheduled for treatment with cytotoxic chemotherapy (Gemcitabine HCL/Carboplatin)
3. Preserved major organ functions, i.e:

   * B-Leukocyte count ≥ 3.0 x 109/L
   * B-Neutrophil count ≥ 1.5 x 109/L
   * B-Platelet count ≥ 75 x109/L
   * B-Haemoglobin ≥ 100 g/L (transfusions are allowed)
   * P-Total bilirubin level ≤ 1.5 times the upper institutional limit of the "normal" (i.e. reference)range
   * P-ASAT or P-ALAT ≤ 2.5 times upper institutional limit of the "normal" range, ≤5 times if liver metastases have been documented
   * P-Creatinine ≤ 1.5 times upper institutional limit of the "normal" range
   * 12-lead ECG with normal tracings; or clinically nonsignificant changes that did not require medical intervention
4. Signed written informed consent.

Exclusion Criteria:

* The presence of any of the following criteria will exclude the patient from participating in the study:

  * Ongoing infection or other major recent or ongoing disease that, according to the investigator, poses an unacceptable risk to the patient
  * Grade 3 or higher constipation within the past 28 days or grade 2 constipation within the past 14 days before randomization. (Patients with grade 2 constipation within the past 14 days could be re-screened if constipation decreases to ≤ grade 1 with optimal management of constipation.)
  * Known malignancy in Central Nervous System (CNS)
  * Disease and dementia and neuropathy grade more than 1
  * Other active malignancy during the previous 3 years
  * Major surgical procedure within 4 weeks
  * Prior anti-tumor therapy apart from radiation therapy
  * Women Of Child Bearing Potential (WOCBP) - For purposes of this study, WOCBP include any female who has experienced menarche and who is not postmenopausal. Post menopause is defined as: Amenorrhea ≥ 12 consecutive months without another cause
  * Pregnancy or lactation
  * Current participation in any other interventional clinical trial
  * Performance status > ECOG 2 after optimization of analgesics
  * Life expectancy less than 3 months
  * Contraindications to the investigational product, e.g. known or suspected hypersensitivity.
  * Lack of suitability for participation in the trial, for any reason, as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety of AXL1717 in combination with Gemcitabine HCL and Carboplatin | End of two cycles, i.e. 6 weeks
  A dose finding pilot study to evaluate safety and pharmacokinetics in combination with Gemcitabine HCL and Carboplatin during two treatment cycles, i.e. 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bergqvist, M.D., Ph.D, Principal Investigator — Uppsala University Hospital, Sweden
Locations (2):
- Sweden (2):
  - KFUE, Uppsala
  - University Hospital, Uppsala